CLINICAL TRIAL: NCT06973174
Title: Bacillus Cereus Invasive Infections in Preterm Neonates Hospitalized in French Hospitals
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 25LaboBacterio01
Record Dates: First submitted 2025-05-05; First posted 2025-05-15 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Sepsis; Infections
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Only the bacteial strains (isolated from patients blood culture samples were retained. Only bacterial DNA was extractable from these samples and not patient DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Premature neonates with invasive infection caused by Bacillus cereus — The whole genome sequencing of the bacterial strains was performed by using both Illumina and Nanopore technologies, allowing us to obatin high quality and complete circular genomes.
  Other Names: Bacterial species identification by Whole Genome sequencing

SUMMARY:
Background. Bacillus cereus group (Bc) comprises twenty-six closely related species of spore-forming environmental bacteria. Recently, increased sepsis and septic shock caused by Bc were reported in preterm neonates (PN), and the mortality rate can reach up to 30%. Using Whole Genome Sequencing (WGS) increasingly used to characterize Bc strains, The team aimed to determine an accurate identification to the species level of the strains involved in Bc invasive infections in preterm neonates in France and study their virulome profile.Methods. The team performed WGS for 40 neonate clinical strains responsible for invasive infections in PN. A screening of virulence genes was performed to characterize strains associated with poor prognosis. Clinical data were collected and all clinical and genomic findings were analyzed for risk factors for death.

"

ELIGIBILITY:
Inclusion Criteria:

* Premature newborn (i.e born before 37 last menstrual periods) with invasive infection caused by B. cereus (strains isolated from blood culture and cerebrsopinal fluid)

Exclusion Criteria:

* None

Max Age: 143 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The premature newborn included in the study were recruited from 14 NICU in 14 Tertiary Care center in France. This study is a national retrospective study
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-01-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days after birth
  The mortality at D28 after birth was collected in patients record.

CONTACTS AND LOCATIONS:
Locations (13):
- France (13):
  - CHU NICE, Nice, Alpes Maritimes
  - CHU lille, Lille
  - AP-HM Marseille, Marseille
  - CHU Nantes, Nantes
  - CHU Nîmes, Nîmes
  - AP-HP Hôpital Robert Debré, Paris
  - Hôpital Antoine Béclère, AP-HP, Paris
  - Hôpital Cochin, Paris
  - CHU de Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHRU de Strasbourg, Strasbourg
  - CHU Toulouse, Toulouse
  - CHU de Tours, Tours